CLINICAL TRIAL: NCT02789280
Title: Mood Management Effects of Brief Unsupported Internet Interventions
Brief Title: Mood Management Effects of Brief Unsupported Internet Interventions II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i4Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-009 - H Part II
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-04

CONDITIONS: Mood
MeSH Terms: interventions — Exercise; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activities. (Experimental): Increasing activity level included a brief description of how activities affect mood. Participants were then asked to choose the activities they could use to improve their mood from an available list of "helpful activities"; users were also able to generate their own helpful activities. Participants were also presented with examples of unhelpful activities such as staying in bed and being isolated.
  Interventions: Behavioral: Activities.
- Wait List (Active Comparator): Participants will be asked to wait for a week until they receive the behavioral activation condition
  Interventions: Other: Wait list

INTERVENTIONS:
Behavioral: Activities. — Increasing activity level included a brief description of how activities affect mood. Participants were then asked to choose the activities they could use to improve their mood from an available list of "helpful activities"; users were also able to generate their own helpful activities. Participants were also presented with examples of unhelpful activities such as staying in bed and being isolated
  Arms: Activities.
Other: Wait list — will receive the behavioral activation condition after one week of completing baseline assessment.
  Arms: Wait List

SUMMARY:
The main goal of this study was to compare the effect of a one-session unsupported Internet intervention on participants' clinical symptoms (depressive and anxiety symptoms) and related variables (mood, confidence and motivation).

DETAILED DESCRIPTION:
The main goal of this study was to compare the effect of a one-session unsupported Internet intervention on participants' clinical symptoms (depressive and anxiety symptoms) and related variables (mood, confidence and motivation).

Method: A total of 275 adults residing in the United States will take part in a randomized controlled trial. Participants were randomly assigned to an experimental condition based on Behavioral activation or a one week wait list condition. They will be follow-up one week after consenting.

ELIGIBILITY:
Inclusion Criteria:

* most be U.S. citizens

Exclusion Criteria:

* non-U.S. residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9; Kroenke & Spitzer, 2002) scores | Baseline - 1 week follow-up
  Which is a widely used 10-item measure that screens for a presence of a major depressive episode as well as assesses the severity of depressive symptomatology over a 2-week period.

SECONDARY OUTCOMES:
Mood- Likert-type question | Baseline - 10 minutes after the intervention - 1 week follow-up
  How would you describe your mood in the last 2 weeks? and had responses ranging from 0 = Extremely Negative to 9 = Extremely Positive
Motivation - Likert-type question | Baseline - 10 minutes after the intervention - 1 week follow-up
  How motivated are you to do something to improve your mood? and had responses ranging from 0 = Extremely Negative to 9 = Extremely Positive
Confidence - Likert-type question | Baseline - 10 minutes after the intervention - 1 week follow-up
  How confident are you that you are able to do something to improve your mood?and had responses ranging from 0 = Extremely Negative to 9 = Extremely Positive
Usefulness - Likert-type question | Baseline - 10 minutes after the intervention
  Before you see the ideas we will be sharing with you, how likely do you think they will be useful?" and had responses ranging from 0 = Very Unlikely to 6 = Very Likely.
7-item Generalized Anxiety Disorder questionnaire | Baseline - 1 week follow-up
  self-report questionnaire for measuring the level of generalized anxiety symptoms over a two-week period

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Muñoz, Ph.D, Principal Investigator — Palo Alto University
Locations (1):
- Palo Alto University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No